CLINICAL TRIAL: NCT02743897
Title: Open-Labeled Trial Of Direct-Acting Antiviral Treatment Of Hepatitis C-Negative Patients Who Receive Kidney Transplants From Hepatitis C-Positive Donors
Brief Title: Transplanting Hepatitis C Kidneys Into Negative Kidney Recipients
Acronym: THINKER
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 823833
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: End Stage Renal Disease
Keywords: end-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — elbasvir-grazoprevir drug combination; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Direct-acting antiviral treatment for HCV (Experimental)
  Interventions: Drug: Zepatier; Drug: Mavyret

INTERVENTIONS:
Drug: Zepatier — Zepatier (grazoprevir 100mg and elbasvir 50 mg once daily) is taken by mouth for 12 weeks unless a genetic variation is detected. In this case treatment with Zepatier will be extended to 16 weeks. Study subjects with treatment failure will be provided open-label Zepatier + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.
Drug: Mavyret — Mavyret (glecaprevir 100 mg and pibrentasvir 40 mg) is taken by mouth for 8 weeks. Study subjects with treatment failure will be provided an alternative DAA + sofosbuvir (sovaldi) 400mg + Ribavirin (generic), renally dosed based on creatinine clearance per the manufacturer guidelines.

SUMMARY:
This study is being conducted to determine safety and effectiveness of transplanting kidneys from Hepatitis C-positive donors into Hepatitis C-negative patients on the kidney transplant waitlist, who will then be treated with the appropriate direct-acting antiviral (DAA) after the single kidney transplantation.

DETAILED DESCRIPTION:
Open-labelled pilot clinical trial of Zepatier (Grazoprevir + Elbasvir), Mavyret (Glecaprevir + Pibrentasvir), Epclusa (Sofosbuvir + Velpatasvir), or another appropriate DAA in at least 75 HCV-negative subjects with end-stage renal disease receiving a kidney transplant from a HCV-positive donor. Eligible subjects will receive a kidney transplant from a deceased-donor, and then will receive DAA treatment after kidney transplantation when infection with HCV is confirmed in these kidney transplant recipients. Treatment will be complete after 12 weeks for most subjects.

ELIGIBILITY:
Subject:

Inclusion criteria

* Must be waitlisted for a kidney transplant (dialysis is not a requirement if a patient is waitlisted)
* Listed for an isolated kidney transplant with ≤2555 days of accrued transplant waiting time and/or ≤2555 days of dialysis time for blood group A, B, or O, by enrollment
* Listed for an isolated kidney transplant with ≤1825 days of accrued transplant waiting time and/or ≤1825 days of dialysis time for blood group AB, by enrollment
* No available living kidney donor
* Between 30-70 years of age, by enrollment
* Have a panel reactive antibody level ≤97%
* eGFR <15ml/min/1.73m2 as calculated using the 4 variable MDRD equation
* Obtained agreement for participation from the patient's treating transplant nephrologist
* Able to travel to the University of Pennsylvania for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
* No active illicit substance abuse
* Weigh at least 50kg
* Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant due to the increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method to prevent any secretion exchange
* Inclusion criteria for treatment (not for entry as study patient) will include any detectable HCV RNA
* Able to provide informed consent

Exclusion criteria

* Hepatocellular carcinoma
* Patients with primary focal segmental glomerulosclerosis (FSGS), FSGS recurring after previous transplant, or disease process with increased risk of causing early graft failure as per the treating nephrologist
* HIV positive
* HCV RNA positive (can be isolated HCV antibody positive provided the subject has no history of previously treated HCV)
* Hepatitis B surface antigen positive
* Any other chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD) with abnormal liver enzymes
* Persistently elevated liver transaminases
* Significant hepatic fibrosis on screening elastography (≥f2 fibrosis)
* Pregnant or nursing (lactating) women
* Known allergy or intolerance to tacrolimus that would require post-transplant administration of cyclosporine, rather than tacrolimus given the drug-drug interaction between cyclosporine and Zepatier
* Waitlisted for a multi-organ transplant (e.g., pancreas-kidney, heart-kidney, etc.)
* Significant cardiomyopathy defined as either:

  * Left ventricular ejection fraction <40% on most recent echocardiogram
  * Left ventricular ejection fraction ≥40% but <50% on most recent echocardiogram with an <5 METS of exercise tolerance
  * Reversible ischemia on stress testing without revascularization

Donor Organ Selection:

Inclusion Criteria

* Detectable HCV RNA
* Age ≤60 years
* Study modified Kidney donor profile index (KDPI) score ≤0.856 - calculated as if the kidney were HCV-negative (https://optn.transplant.hrsa.gov/resources/allocation-calculators/kdpi-calculator/)

Exclusion Criteria

* Anatomical issues in the kidney allograft that raise the risk of post-transplant complications (e.g., number or length of renal arteries or veins)
* Confirmed HIV positive
* Confirmed HBV positive (positive Hepatitis B surface antigen and/or HBV DNA)
* Known previously failed treatment for HCV using a regimen with a direct-acting antiviral (can have received interferon monotherapy and/or interferon + ribavirin combination therapy)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Prenner, MD, Principal Investigator — University of Hospital of Pennsylvania; Peter Reese, MD, MSCE, Principal Investigator — University of Hospital of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sulkowski M, Hezode C, Gerstoft J, Vierling JM, Mallolas J, Pol S, Kugelmas M, Murillo A, Weis N, Nahass R, Shibolet O, Serfaty L, Bourliere M, DeJesus E, Zuckerman E, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 8 weeks versus 12 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin in patients with hepatitis C virus genotype 1 mono-infection and HIV/hepatitis C virus co-infection (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1087-97. doi: 10.1016/S0140-6736(14)61793-1. Epub 2014 Nov 11. PMID 25467560
- [Background] Lawitz E, Gane E, Pearlman B, Tam E, Ghesquiere W, Guyader D, Alric L, Bronowicki JP, Lester L, Sievert W, Ghalib R, Balart L, Sund F, Lagging M, Dutko F, Shaughnessy M, Hwang P, Howe AY, Wahl J, Robertson M, Barr E, Haber B. Efficacy and safety of 12 weeks versus 18 weeks of treatment with grazoprevir (MK-5172) and elbasvir (MK-8742) with or without ribavirin for hepatitis C virus genotype 1 infection in previously untreated patients with cirrhosis and patients with previous null response with or without cirrhosis (C-WORTHY): a randomised, open-label phase 2 trial. Lancet. 2015 Mar 21;385(9973):1075-86. doi: 10.1016/S0140-6736(14)61795-5. Epub 2014 Nov 11. PMID 25467591
- [Background] Forns X, Gordon SC, Zuckerman E, Lawitz E, Calleja JL, Hofer H, Gilbert C, Palcza J, Howe AY, DiNubile MJ, Robertson MN, Wahl J, Barr E, Buti M. Grazoprevir and elbasvir plus ribavirin for chronic HCV genotype-1 infection after failure of combination therapy containing a direct-acting antiviral agent. J Hepatol. 2015 Sep;63(3):564-72. doi: 10.1016/j.jhep.2015.04.009. Epub 2015 Apr 18. PMID 25895428
- [Background] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356
- [Background] O'Leary JG, Neri MA, Trotter JF, Davis GL, Klintmalm GB. Utilization of hepatitis C antibody-positive livers: genotype dominance is virally determined. Transpl Int. 2012 Aug;25(8):825-9. doi: 10.1111/j.1432-2277.2012.01498.x. Epub 2012 May 30. PMID 22643162
- [Background] Roth D, Nelson DR, Bruchfeld A, Liapakis A, Silva M, Monsour H Jr, Martin P, Pol S, Londono MC, Hassanein T, Zamor PJ, Zuckerman E, Wan S, Jackson B, Nguyen BY, Robertson M, Barr E, Wahl J, Greaves W. Grazoprevir plus elbasvir in treatment-naive and treatment-experienced patients with hepatitis C virus genotype 1 infection and stage 4-5 chronic kidney disease (the C-SURFER study): a combination phase 3 study. Lancet. 2015 Oct 17;386(10003):1537-45. doi: 10.1016/S0140-6736(15)00349-9. Epub 2015 Oct 5. PMID 26456905
- [Background] Reese PP, Abt PL, Blumberg EA, Goldberg DS. Transplanting Hepatitis C-Positive Kidneys. N Engl J Med. 2015 Jul 23;373(4):303-5. doi: 10.1056/NEJMp1505074. No abstract available. PMID 26200976
- [Background] Reddy KR FS, et al. Ledipasvir/Sofosbuvir with Ribavirin for the Treatment of HCV in Patients with Post Transplant Recurrence: Preliminary Results of a Prospective, Multicenter Study. Hepatology. 2014;60:200A
- [Background] Van Deerlin, V. (December 2015). Hepatitis C Virus Genotyping (GenMark Assay) Validation Summary
- [Background] Pawlak R RJ, Maranan G, Michel-Treil V, Schutzbank T. A Comparative Evaluation of the Siemens VERSANT HCV Genotype 2.0 (LiPA) and GenMark eSensor HCV Direct Genotyping Tests. CVS 2013 Covance; 2013
- [Background] Dahl A HD, Ogorek T, Hansen G. Comparison of the GenMark Direct Genotype Assay with the LiPA Genotype Assay Using a Diverse Spectrum of HCV Clinical Samples Encountered in a High Risk Inner City HCV Population. CVS 2013 Hennepin; 2013.
- [Background] Woodberry M SK, Castor J, Cook L, Jerome K. Genotyping of Hepatitis C Virus by the Genmark DX Esensor HCVG Direct Test. CVS 2013 UW-Seattle 2013
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Cancer Institute. (June 2010). Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
- [Background] Merck Sharp & Dohme Corporation (January 2016). ZEPATIER™ tablets. Highlights of Prescribing Information. 2016.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Elbasvir (MK-8742). Investigator's Brochure (8th Ed.). 2015.
- [Background] Merck Sharp & Dohme Corporation (July 2015). Grazoprevir (MK-5172). Investigator's Brochure (10th Ed.). 2015.
- [Derived] Sawinski D, Forde KA, Lo Re V 3rd, Goldberg DS, Cohen JB, Locke JE, Bloom RD, Brensinger C, Weldon J, Shults J, Reese PP. Mortality and Kidney Transplantation Outcomes Among Hepatitis C Virus-Seropositive Maintenance Dialysis Patients: A Retrospective Cohort Study. Am J Kidney Dis. 2019 Jun;73(6):815-826. doi: 10.1053/j.ajkd.2018.11.009. Epub 2019 Jan 29. PMID 30704882
- [Derived] Reese PP, Abt PL, Blumberg EA, Van Deerlin VM, Bloom RD, Potluri VS, Levine M, Porrett P, Sawinski D, Nazarian SM, Naji A, Hasz R, Suplee L, Trofe-Clark J, Sicilia A, McCauley M, Gentile C, Smith J, Niknam BA, Bleicher M, Reddy KR, Goldberg DS. Twelve-Month Outcomes After Transplant of Hepatitis C-Infected Kidneys Into Uninfected Recipients: A Single-Group Trial. Ann Intern Med. 2018 Sep 4;169(5):273-281. doi: 10.7326/M18-0749. Epub 2018 Aug 7. PMID 30083748
- See also: Quest Diagnostics, Inc. (December 2014). Test summary guide. Hepatitis C Viral RNA Genotype 1 NS5a Drug Resistance. — http://www.questdiagnostics.com/testcenter/testguide.action?dc=TS_HCV_NS5A_Genotype&tabview=true
- See also: Sandoz, Inc. (May 2015) Ribavirin capsule. Highlights of Prescribing Information. 2015. — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?setid=dc637c8f-9669-4bc5-8787-1fd5abaa588e.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct-acting Antiviral Treatment for HCV
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 62
Age, Customized [Median (Inter-Quartile Range); unit: years] | 57 [50 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 29
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Cured
Description: Subjects with post-treatment sustained virologic response (SVR) = Number of subjects with negative HCV RNA 12 weeks after completing therapy / number of subjects treated post-kidney transplantation
Time Frame: Baseline to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 62
Participants | 62

2. Primary Outcome: Number of Subjects With SAE Attributable to HCV Therapy
Description: Number of subjects with major adverse events attributable to HCV therapy in post-kidney transplant
Time Frame: Baseline to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Direct-acting Antiviral Treatment for HCV
Number analyzed (Participants) | 62
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year post-transplant
Arm/Group | Direct-acting Antiviral Treatment for HCV
All-Cause Mortality (participants affected / at risk) | 1/62
Serious Adverse Events (participants affected / at risk) | 2/62
Other Adverse Events (participants affected / at risk) | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Direct-acting Antiviral Treatment for HCV (N=62)
Focal segmental glomerulosclerosis (FSGS) (Renal and urinary disorders) | 1
Death (Respiratory, thoracic and mediastinal disorders) | 1 — COVID-19 (coronavirus disease)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT02743897/Prot_SAP_000.pdf